CLINICAL TRIAL: NCT05274893
Title: A Randomized, Open-label, Two-cycle Crossover Pharmacokinetic Comparison Study of SYHX2011 and Abraxane® in Patients With Advanced Breast Cancer
Brief Title: A Pharmacokinetic Comparison Study of SYHX2011 and Abraxane® in Patients With Advanced Breast Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SYHX2011-001
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SYHX2011(T)-Abraxane®(R) (Experimental): Patients will be administrated with SYHX2011 followed by Abraxane®
  Interventions: Drug: SYHX2011 and Abraxane®
- Abraxane®(R)-SYHX2011(T) (Experimental): Patients will be administrated with Abraxane® followed by SYHX2011
  Interventions: Drug: SYHX2011 and Abraxane®

INTERVENTIONS:
Drug: SYHX2011 and Abraxane® — IV infusion, 260 mg/m^2

SUMMARY:
This is a multi-center, open-label, pharmacokinetic comparison study of SYHX2011 and Abraxane® in patients with advanced breast cancers after single IV infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the written informed consent.
2. Female patients aged 18 to 75 years (inclusive).
3. Histologically and/or cytologically diagnosed advanced breast cancer.
4. Patients who are receiving paclitaxel for injection (albumin bound) monotherapy or who, in the judgement of the investigator, may benefit from monotherapy with the trial formulation.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
6. Expected survival time ≥3 months.
7. The results of hematological, renal, and hepatic function are within the following ranges:

   White blood cell count (WBC) ≥3.0 × 10^9/L; Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L; Platelet count (PLT)≥ 100 × 10^9/L; Hemoglobin (Hb) ≥ 90 g/L; Prothrombin time (PT)/activated partial thrombin time (APTT) ≤1.5 × ULN; Total bilirubin (TBIL) ≤ 1.5 × ULN; AST、ALT ≤ 2.5 × ULN (≤5 × ULN in patients with liver metastasis); Serum creatinine ≤ 1.5 × ULN.
8. Patients have no pregnancy plan within 6 months after entering the study, voluntarily take effective contraceptive measures, and have no egg donation plan.
9. Fully understand the purpose and requirements of this trial, and can complete the whole trial process according to the test requirements.

Exclusion Criteria:

1. Have severe allergy to paclitaxel drugs or human serum albumin, or history of significant hypersensitivity or idiosyncratic reaction.
2. Patients with serious medical conditions are considered unsuitable for inclusion by the investigator.
3. Patients who have undergone major surgery within 3 months prior to screening or planned to have major surgery during the study period.
4. Have a history of alcohol, drug abuse or drug addiction.
5. Patients who are pregnant or breasting.
6. Patients with one or more positive tests for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), human immunodeficiency virus (HIV) or treponema pallidum antibody.
7. Received anti-tumor therapy such as radiotherapy, biotherapy, endocrine therapy, targeted therapy, immunotherapy, chemotherapy [paclitaxel for injection (albumin bound) monotherapy less than 21 days] within 4 weeks prior to study dosing or participated in other clinical trials within the 5 half-lives of the treated drug, whichever is longer. According to the determination of the investigator, the washout period can be appropriately shortened or extended. If there are interfering monoclonal antibodies that require an appropriate extension of the washout period when necessary, or if other antitumor drugs need to be combined during the study.
8. Obvious abnormality in ECG examination, QTc interval > 470 ms at baseline.
9. Peripheral neuropathy ≥ grade 2.
10. Blood donation or massive blood loss (> 400 mL) within 90 days before screening.
11. Use of drugs with high protein binding rate, or CYP2C8 inhibitors, or CYP3A4 inhibitors, within 1 week before enrollment.
12. Ingestion of a specific diet (e.g., grapefruit) within 48 hours prior to the administration of the study drug, capable of affecting the absorption, distribution, metabolism, and excretion of the drug.
13. Toxicity due to antitumor drug use before enrollment did not recover to ≤ grade 1 or baseline, except for alopecia.
14. Not suitable for this study as judged by the investigator for any other reason.

    -

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-03-31 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Cmax | From time zero up to 72 hours post-dose
  Maximum plasma concentration
AUC0-t | From time zero up to 72 hours post-dose
  Area under the plasma concentration time curve from time zero to the last measurable concentration
AUC0-∞ | From time zero up to 72 hours post-dose
  Area under the plasma concentration-time curve from time zero to infinity

CONTACTS AND LOCATIONS:
Overall Officials: Mingxia Wang, Principal Investigator — Hebei Medical University Fourth Hospital

IPD SHARING:
Plan to Share IPD: No